CLINICAL TRIAL: NCT01981499
Title: A Phase 1, Placebo-Controlled, Crossover, Subject- And Investigator-Blind, Sponsor-Open Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Effects On Histamine-Induced Wheal Of A Modified-Release Formulation Of PF-05180999 In Healthy Adult Subjects
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, And Effects On Histamine-Induced Wheal Of PF-05180999 In Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was prematurely terminated on 01April2014 due to safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B3441009
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Migraine
Keywords: PF-05180999; safety; tolerability; pharmacokinetics; histamine; wheal; flare; migraine; PDE2
MeSH Terms: conditions — Migraine Disorders; Urticaria | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm A1 (Experimental): Part A of study to assess safety, tolerability, and pharmacokinetics of PF-05180999
  Interventions: Drug: PF-05180999
- Arm A2 (Placebo Comparator): Part A of study to assess safety, tolerability, and pharmacokinetics of PF-05180999 relative to placebo
  Interventions: Drug: Placebo
- Arm B1 (Experimental): Part B of study to assess effects of PF-05180999 on histamine-induced wheal
  Interventions: Drug: 120 mg MR PF-05180999
- Arm B2 (Experimental): Part B of study to assess effects of PF-05180999 on histamine-induced wheal
  Interventions: Drug: 360 mg MR PF-05180999
- Arm B3 (Experimental): Positive control to ensure histamine-induced wheal assay integrity
  Interventions: Drug: 10 mg cetirizine
- Arm B4 (Experimental): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05180999 — Ascending single oral doses of 120, 240, and 420 mg modified-release tablets
  Arms: Arm A1
Drug: Placebo — Placebo tablets
  Arms: Arm A2
Drug: 120 mg MR PF-05180999 — Single 120 mg dose administered as modified release formulation
  Arms: Arm B1
Drug: 360 mg MR PF-05180999 — Single 360 mg dose administered as modified release formulation
  Arms: Arm B2
Drug: 10 mg cetirizine — Single 10 mg dose of cetirizine
  Arms: Arm B3
Drug: Placebo — Placebo tablets
  Arms: Arm B4

SUMMARY:
PF-05180999 is a phosphodiesterase-2 inhibitor that is hypothesized to be able to reduce vascular permeability. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and effects on histamine-induced wheal of single doses of PF-05180999 in healthy adult subjects. Histamine-induced wheals are biomarkers of vascular permeability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years
* No history of clinically-relevant atopic or dermatological disease
* Positive reaction to intradermal injection of histamine

Exclusion Criteria:

* Subjects with screening laboratory test results that deviate from the upper and/or lower limits of the reference or acceptable range. The exception is that all liver function tests must not exceed the upper limit of normal.
* Subjects with evidence of, or history of, hepatic disorder, including acute or chronic hepatitis B or hepatitis C
* Intolerance to intradermal histamine injection.
* Subjects with dark skin (Part B only).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0-72 hours post-dose
  Maximum observed plasma concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-72 hours post-dose
  Time when Cmax occurred
Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-72 hours post-dose
  Measure of drug absorption and drug exposure
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) | 0-infinity hours post-dose
  Measure of drug absorption and drug exposure
Plasma Half-Life (t1/2) | 0-72 hours post-dose
  Time for the plasma concentration to decrease by one-half.
Area Under the Effect Curve (AUEC) for Histamine-Induced Wheal | 2-12 hours post-dose
  Measure of drug effect

SECONDARY OUTCOMES:
Dose-response, exposure-response, and maximum response for PF-05180999 against histamine-induced wheal | 0-72 hours post-dose
  Measures of drug effect
Area Under the Effect Curve (AUEC) for histamine-induced flare; Dose-response, exposure-response, and maximum response for PF-05180999 against histamine-induced flare | 0-72 hours post-dose
  Measures of drug effect

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Saint Paul, Minnesota, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3441009&StudyName=A%20Study%20of%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Effects%20On%20Histamine-Induced%20Wheal%20Of%20PF-05180999%20In%20Healthy%20Adults%20%20